CLINICAL TRIAL: NCT03590938
Title: Lynparza Tablets 100mg, 150mg CEI, Investigation on Development of Bone Marrow Depression in Patients With Unresectable or Recurrent BRCA Mutated HER2 Negative Breast Cancer Who Have Previously Received Anticancer Chemotherapy
Brief Title: Lynparza Breast Cancer Clinical Experience Investigation
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D0819C00005
Record Dates: First submitted 2018-06-27; First posted 2018-07-18 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To characterise the development of ADRs of bone marrow depression in patients under actual post-marketing use

DETAILED DESCRIPTION:
To characterise the development of adverse drug reactions (ADRs) of bone marrow depression in patients with unresectable or recurrent BRCA mutated HER2 negative breast cancer who have previously received anticancer chemotherapy under actual post-marketing use.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable or recurrent BRCA mutated HER2 negative breast cancer with prior anticancer chemotherapy

Exclusion Criteria:

* The patients who are not started on Lymparza for the first time

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Investigation sites mainly consisted of department of surgical related department (surgery, mammary gland surgery, and endocrine surgery, etc.) and department of internal medicine.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
Adverse drug reactions of bone marrow depression | One year period
  Bone marrow depression will be investigated as safety specification topics

CONTACTS AND LOCATIONS:
Overall Officials: Toshimitsu Tokimoto, Study Director — AstraZeneca KK
Locations (31):
- Japan (31):
  - Research Site, Aichi
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukui
  - Research Site, Fukuoka
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Ishikawa
  - Research Site, Kagawa
  - Research Site, Kagoshima
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kyoto
  - Research Site, Miyagi
  - Research Site, Nagano
  - Research Site, Nara
  - Research Site, Okayama
  - Research Site, Okinawa
  - Research Site, Osaka
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shimane
  - Research Site, Shizuoka
  - Research Site, Tokyo
  - Research Site, Toyama
  - Research Site, Yamagata
  - Research Site, Yamaguchi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0819C00005&attachmentIdentifier=d8a01299-bcfa-4ad7-9c00-c66ca8ff52d6&fileName=D0819C00005-Synopsis.pdf&versionIdentifier=